CLINICAL TRIAL: NCT02633137
Title: Sequential Chemotherapy and Lenalidomide Followed by Rituximab and Lenalidomide Maintenance for Untreated Mantle Cell Lymphoma: A Phase II Study
Brief Title: Sequential Chemotherapy and Lenalidomide Followed by Rituximab and Lenalidomide Maintenance for Untreated Mantle Cell Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Celgene Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15-196
Record Dates: First submitted 2015-12-15; First posted 2015-12-17 (Estimated); Results first posted 2024-08-30 (Actual); Last update posted 2024-08-30 (Actual); Status verified 2023-11

CONDITIONS: Mantle Cell Lymphoma; Untreated
Keywords: Lenalidomide; 15-196
MeSH Terms: conditions — Lymphoma, Mantle-Cell | interventions — Lenalidomide; R-CHOP protocol; Cytarabine

ARMS (1):
- Chemotherapy (Experimental): Lenalidomide + R-CHOP x 4 cycles R-HiDAC x 2 cycles R-Len maintenance x 6 months. Patients will be followed on active follow up for three years after completion of therapy. After the active followup period, survival, relapse, and new anti-lymphoma therapy information will be collected via telephone calls, patient medical records, and/or clinic visits approximately every 6 months until death, loss to follow up or consent withdrawal, whichever comes first.
  Interventions: Drug: Lenalidomide; Drug: R-CHOP; Drug: high-dose cytarabine (HIDAC)

INTERVENTIONS:
Drug: Lenalidomide
Drug: R-CHOP — * Rituximab 375 mg/m^2 IVPB with premedications Day 1
  * Cyclophosphamide 750 mg/m^2 IVPB Day 1
  * Doxorubicin 50 mg/m^2 IVP Day 1
  * Vincristine 1.4 mg/m^2 IVP (capped at 2 mg) Day 1
  * Prednisone 100 mg PO Daily on Days 1-5 or 2-6
Drug: high-dose cytarabine (HIDAC)

SUMMARY:
The purpose of this study is to find out what effects, good and/or bad, the treatment including 1) Lenalidomide-RCHOP, 2) R-HIDAC, and 3) Lenalidomide-Rituximab maintenance has on the participant and their lymphoma.

DETAILED DESCRIPTION:
Patients will receive lenalidomide 15 mg orally daily on days 1-14 with standard-dose R-CHOP (375 mg/m^2 intravenous rituximab, 750 mg/m2 intravenous cyclophosphamide, 50 mg/m^2 intravenous doxorubicin, and 1.4 mg/m2 intravenous vincristine on day 1, and 100 mg prednisone days 1-5 or days 2-6) every 21 days for four cycles.

All patients will receive pegfilgrastim on day 2 of each cycle and aspirin 81 mg orally daily for venous thromboembolism prophylaxis throughout the four cycles.

After four cycles of Len-RCHOP, the patients will undergo restaging PET/CT scans. Patients with evidence of disease progression will be treated off study.

R-HIDAC After lenalidomide-RCHOP phase, patients without evidence of progressive disease will receive rituximab 375 mg/m^2 day 1 and then patients will be admitted for high-dose cytarabine (HIDAC). Recommended age-adjusted HIDAC doses are as follows: ≤65 years: 3 g/m2 every12 hours X 4 doses; 65-70 years: 2 g/m^2 every12 hours X 4 doses; >70 years: 1 g/m^2 every12 hours X 4 doses. Physician discretion will dictate the choice of HIDAC dose, ranging from 1 g/m^2 - 3 g/m^2 every 12 hours X 4 doses.

Patients will receive two cycles of rituximab-HIDAC every 3 weeks. After two cycles of R-HIDAC, the patients will undergo restaging PET/CT scans. Patients with evidence of disease progression will be treated off study.

Len-Rituximab Maintenance After completion of induction chemotherapy with Len-RCHOP and R-HIDAC, patients will begin maintenance phase with lenalidomide and rituximab for 6 months. Lenalidomide will be administered at 15 mg orally daily on days 1-21 of a 28-day cycle for a total of 6 cycles and rituximab maintenance every 8 weeks for a total of 3 treatments.

ELIGIBILITY:
Inclusion Criteria:

* Previously untreated mantle cell lymphoma patients (at least clinical stage 2)
* Histologic diagnosis confirmed by MSKCC pathologist as mantle cell lymphoma
* Presence of evaluable disease
* Age ≥18 years KPS ≥ 70%
* Adequate organ function: ANC ≥1500 and platelet count ≥100,000, unless felt to be secondary to underlying mantle cell lymphoma
* Renal function assessed by calculated creatinine clearance as follows:
* Cockcroft-Gault estimation of CrCl):

  * Calculated creatinine clearance ≥ 30ml/min by Cockcroft-Gault formula. See section below, "Dosing Regimen", regarding lenalidomide dose adjustment for calculated creatinine clearance ≥30ml/min and < 60ml/min.
* Adequate hepatic function as determined by

  * Total bilirubin <1.5X upper limit of normal (ULN) (unless known Gilbert syndrome)
  * AST (SGOT) and ALT (SGPT) 3 x ULN
* All study participants must be registered into the mandatory Revlimid REMS® program, and be willing and able to comply with the requirements of the REMS® program.
* Females of reproductive potential must adhere to the scheduled pregnancy testing as required in the Revlimid REMS® program.
* Each subject must sign an informed consent form indicating that he or she understand the purpose of and procedures required for the study and are willing to participate.
* Short course systemic corticosteroids is permissible for disease control, improvement of performance status or non-cancer indication if ≤ 10 days and must be discontinued prior to study treatment.

Exclusion Criteria:

* Known central nervous system (CNS) lymphoma
* Uncontrolled or severe cardiovascular disease or left ventricular ejection fraction <50% as determined by echocardiogram or MUGA.
* Any life-threatening illness, medical condition, or organ system dysfunction which, in the investigator's opinion, could compromise the subject's safety or put the study outcomes at undue risk.
* Pregnant or breast-feeding. Pre-menopausal patients must have a negative serum HCG within 14 days of enrollment.
* Patients using ≥20 mg/day of prednisone (or steroid equivalent dose) for any chronic medical condition
* Known seropositive, requiring anti-viral therapy, and with detectable viral load by PCR for human immunodeficiency virus (HIV), hepatitis B virus (HBV) or hepatitis C virus (HCV).
* Known hypersensitivity to thalidomide or lenalidomide
* The development of erythema nodosum if characterized by a desquamating rash while taking thalidomide or similar drugs.
* Patients planned for upfront consolidation with high-dose therapy and autologous stem cell transplant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2015-12-14; Primary Completion 2023-11-07 (Actual); Study Completion 2023-11-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anita Kumar, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (7):
  - Memorial Sloan Kettering Basking Ridge, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth, Middletown, New Jersey
  - Memorial Sloan Kettering Bergen, Montvale, New Jersey
  - Memorial Sloan Kettering Commack, Commack, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Nassau, Uniondale, New York

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — https://www.mskcc.org/

RESULTS

PARTICIPANT FLOW:
Groups:
- Chemotherapy: Lenalidomide + R-CHOP x 4 cycles R-HiDAC x 2 cycles R-Len maintenance x 6 months.
Period: Overall Study
Arm/Group | Chemotherapy
Started | 49
Completed | 45
Not Completed | 4
Not completed — Adverse Event | 1
Not completed — Lack of Efficacy | 2
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Chemotherapy
Number analyzed (Participants) | 49
Age, Continuous [Median (Full Range); unit: years] | 63 [30 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 36
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 47
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 46
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 49

OUTCOME MEASURES:

1. Primary Outcome: 3-year Progression-free Survival (PFS)
Description: acceptable 3-yr PFS as 75% or higher, and unacceptable rate as 60% or lower.
Time Frame: 3 years
Measure: Number (95% Confidence Interval); unit: % of pts progression-free survival
Arm/Group | Chemotherapy
Number analyzed (Participants) | 49
% of pts progression-free survival | 63 [50 to 78]

ADVERSE EVENTS:
Time Frame: 3 years
Arm/Group | Chemotherapy
All-Cause Mortality (participants affected / at risk) | 18/49
Serious Adverse Events (participants affected / at risk) | 27/49
Other Adverse Events (participants affected / at risk) | 44/49
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Chemotherapy (N=49)
Abdominal pain (Gastrointestinal disorders) | 3
Acute kidney injury (Renal and urinary disorders) | 1
Anemia (Blood and lymphatic system disorders) | 4
Atrial fibrillation (Cardiac disorders) | 3
Other cardiac disorder (Cardiac disorders) | 1
Cholecystitis (Hepatobiliary disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Creatinine increased (Investigations) | 1
Dehydration (Metabolism and nutrition disorders) | 2
Diarrhea (Gastrointestinal disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2
Edema limbs (General disorders) | 1
Enterocolitis infectious (Infections and infestations) | 1
Fatigue (General disorders) | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 23
Fever (General disorders) | 3
Hyponatremia (Metabolism and nutrition disorders) | 1
Other infections and infestations (Infections and infestations) | 1
Joint effusion (Musculoskeletal and connective tissue disorders) | 1
Lung infection (Infections and infestations) | 5
Neutrophil count decreased (Investigations) | 4
Palpitations (Cardiac disorders) | 1
Platelet count decreased (Investigations) | 8
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1
Sepsis (Infections and infestations) | 1
Sinus tachycardia (Cardiac disorders) | 1
Skin infection (Infections and infestations) | 1
Thromboembolic event (Vascular disorders) | 1
Thrombotic thrombocytopenic purpura (Blood and lymphatic system disorders) | 1
Tumor lysis syndrome (Metabolism and nutrition disorders) | 1
White blood cell decreased (Investigations) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Chemotherapy (N=49)
Anemia (Blood and lymphatic system disorders) | 44
Hyperglycemia (Metabolism and nutrition disorders) | 44
Hypoalbuminemia (Metabolism and nutrition disorders) | 40
Neutrophil count decreased (Investigations) | 40
White blood cell decreased (Investigations) | 40
Platelet count decreased (Investigations) | 39
Lymphocyte count decreased (Investigations) | 38
Hypomagnesemia (Metabolism and nutrition disorders) | 21
Alanine aminotransferase increased (Investigations) | 20
Fatigue (General disorders) | 17
Hypocalcemia (Metabolism and nutrition disorders) | 17
Aspartate aminotransferase increased (Investigations) | 16
Alkaline phosphatase increased (Investigations) | 14
Hyperkalemia (Metabolism and nutrition disorders) | 13
Peripheral sensory neuropathy (Nervous system disorders) | 11
Blood bilirubin increased (Investigations) | 10
Constipation (Gastrointestinal disorders) | 10
Hyponatremia (Metabolism and nutrition disorders) | 10
Diarrhea (Gastrointestinal disorders) | 9
Anxiety (Psychiatric disorders) | 7
Back pain (Musculoskeletal and connective tissue disorders) | 7
Creatinine increased (Investigations) | 7
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 7
Hypoglycemia (Metabolism and nutrition disorders) | 7
Hypophosphatemia (Metabolism and nutrition disorders) | 7
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 7
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 7
Arthralgia (Musculoskeletal and connective tissue disorders) | 6
Alopecia (Skin and subcutaneous tissue disorders) | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 5
Edema limbs (General disorders) | 5
Other general disorders and administration site conditions (General disorders) | 5
Hypernatremia (Metabolism and nutrition disorders) | 5
Weight loss (Investigations) | 5
Anorexia (Metabolism and nutrition disorders) | 4
Depression (Psychiatric disorders) | 4
Dizziness (Nervous system disorders) | 4
Hypertension (Vascular disorders) | 4
Myalgia (Musculoskeletal and connective tissue disorders) | 4
Urinary frequency (Renal and urinary disorders) | 4
Activated partial thromboplastin time prolonged (Investigations) | 3
Chest pain-cardiac (Cardiac disorders) | 3
Dry skin (Skin and subcutaneous tissue disorders) | 3
Fever (General disorders) | 3
Headache (Nervous system disorders) | 3
Other infections and infestations (Infections and infestations) | 3
Mucositis oral (Gastrointestinal disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-02-17): https://cdn.clinicaltrials.gov/large-docs/37/NCT02633137/Prot_SAP_000.pdf